CLINICAL TRIAL: NCT06114693
Title: Parameters of the Recovery Time of Acute Kidney Injury in Critically Ill Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed abdelmongy mohamed zayed, Director, Assiut University
Other Study IDs: AKI
Record Dates: First submitted 2023-09-26; First posted 2023-11-02 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-11

CONDITIONS: AKI - Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
the primary objective of this study is to identify and analyze parametrers affecting the time of recovery of AKI in critical ill patient ,Specifically, the study aims to:

1. to identify outcomes of critically ill patients who experienced AKI
2. Examine the relationship between demographic and clinical variables (e.g., age, gender, comorbidities) and outcome of AKI patient
3. follow Baseline characteristics and laboratory findings of the patients at the time of admission to the intensive care unit and affecting it at recovery time
4. Explore the association between psychosocial factors (e.g., depression, anxiety, social support) and outcome of AKI patient at icu

DETAILED DESCRIPTION:
cute kidney injury (AKI) is a common diagnosis in the adult intensive care unit (ICU) due to substantial short- and long-term morbidity and mortality associated with its occurence.AKI globally impacts more than 13 million patients, resulting in approximately 2 million deaths annually.In the United States, it has been estimated that up to 10% of hospi-talizations and up to 60% of patients admitted to an ICU experience AKI. AKI is an abrupt (within hours) decrease in kidney function defined as an increase in serum creatinine (SCr) or a decrease in urine output (UO) for a duration between 7 and 90 days after exposure to an AKI-causing event.The etiology is complex and routinely multifactorial. Known common risk factors associated with AKI inclde diabetes, hypertension, chronic kidney disease (CKD), cardiovascular, lung, and liver diseases, sepsis and surgical interventions, as well as exposure to nephrotoxic medications and diagnostic contrast agents.Despite the development of numerous prevention strategies, the most recent data suggest the incidence of AKI is increasing in the critically ill population.The Kidney Disease Improving Global Outcomes (KDIGO) 2012 workgroup classifies AKI into three stages based on SCr and UO values. AKI is defined within 1week after ICU admission as any of the following: increase in SCr by ⩾0.3mg/dL within 48 h, or increase in SCr to ⩾1.5 times baseline within 1week, or urine output<0.5 mL/kg/hour for 6 h. Severe AKI is defined as KDIGO stage II or stage III AKI .However, SCr and UO measurements remain the standard for evaluation, yet are insensitive and nonspecific markers of AKI and do not account for the etiology or duration of the injury. Despite consensus guidelines for the diagnosis of AKI, discrepancies remain when defining AKI upon ICU admission. Numerous factors influence SCr laboratory measurement such as gender, age, muscle mass, nutritional status, and chronic illness potentially lead-ing to inaccurate estimation of glomerular filtration rate (eGFR). Furthermore, UO can be influenced by a myriad of factors such as effective circulating volume status, hemody-namic status, and medications that impact urinary excretion. Despite current AKI staging guidelines being widely accepted, accuracy of eGFR remains challenging. The strong and independent relationship between AKI and short-term mortality is well described among ICU patients.Short-term outcomes of AKI include alterations in acid-base and electrolyte balance, uremia, and volume overload.Long-term consequences of AKI can be equally devastating and have been associated with acceleration and progression to CKD and end-stage renal disease (ESRD), resulting in the need for lifelong dialysis, renal transplantation, and an exorbitant increase in healthcare expenditures.Therefore, there is a critical need to identify high-risk patients for AKI, the impact of medication use on its incidence, recovery patterns, and clinical outcomes such as mortality, length of stay, and need for mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

1:adult patients (age ≥ 18 years) who admitted to the ICU for at least 24 hours and experience AKI

Exclusion Criteria:

1. patients (age <18 years)
2. Patient who refuse enter study Patient

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients who admitted to the ICU for at least 24 hours and experience AKI
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
parameters as renal arterial resistive index and its effect at recovery time of aki patient at icu | 1year
  comorbidities(DM,HTN,cardiac disease ) sepsis Renal arterial resistive index

IPD SHARING:
Plan to Share IPD: No